CLINICAL TRIAL: NCT04384263
Title: The Influence of Acute and Chronic Tai Chi Practice on Blood Pressure and Brain Health Among Older Adults with Hypertension
Brief Title: The Influence of Tai Chi Practice on Blood Pressure and Brain Health Among Older Adults with Hypertension (ACTION)
Acronym: ACTION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Linda Pescatello, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H19-222; Internal award (Other: UConn)
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Cognitive Decline
Keywords: Tai Chi; Hypertension; Cognitive decline; Brain imaging
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi group (Experimental): During the 12-week online Tai Chi intervention, participants in the Tai Chi group will attend live online Tai Chi sessions led by a certified Tai Chi instructor for 3 sessions/week, 45 minutes/session for 12 weeks. The participants will also practice Tai Chi offline between sessions using instructional videos that will be shared with them at the end of each live online Tai Chi session.
  Participants in the Tai Chi group will be instructed: 1) to maintain their regular level of physical activity outside of the live online Tai Chi exercise sessions and offline Tai Chi exercise, and diet during the study; and 2) to inform the researchers when there is a change(s) in a medical condition or medication prescribed.
  Interventions: Behavioral: Tai Chi
- control (No Intervention): Participants in the control group will perform only their regular habitual daily activities throughout the 12 weeks of intervention period.
  Participants in the control group will be instructed: 1) to maintain their regular level of physical activity and diet during the study; and 2) to inform the researchers when there is a change(s) in a medical condition or medication prescribed.

INTERVENTIONS:
Behavioral: Tai Chi — Participants in the Tai Chi group will practice a Yang style, 8-form Tai Chi routine. Specifically, the routine will incorporate slow, deep breathing and mental relaxation by utilizing Tai Chi movements which: 1) are slow and smooth; 2) without break or pause; and 3) have minimal muscular force and exertion. In addition, investigators will emphasize the breathing techniques of Tai Chi exercise. Investigators will adopt methods of progression to enable the participants learn and safely adapt to the Tai Chi routine and improve skills of practicing, specifically: 1) Tai Chi forms will be taught one at a time; 2) participants will receive instructional videos with step-by-step instructions of how to perform the new Tai Chi form that has been taught in the live online Tai Chi exercise session. Participants will be encouraged to practice Tai Chi offline between live online Tai Chi exercise sessions; however, no time requirement will be proposed.
  Arms: Tai Chi group

SUMMARY:
High blood pressure and poor cognitive function are two common health problems among older adults in the United States. They are also closely related because high blood pressure may lead to negative changes in brain structure and function such as poor brain blood flow that can cause poor cognitive function. Executive function is one type of cognitive function that let people plan and perform difficult tasks. It is commonly damaged by high blood pressure. It is also very important for older adults because they need good executive function to live on their own. Tai Chi is a good exercise option for older adults because it is safe, fun, and social. Research studies show that Tai Chi can reduce blood pressure and improve cognitive function, especially executive function. However, researchers do know if these heart and brain health benefits of Tai Chi are connected.

In the ACTION study, researchers will first measure how a single session of Tai Chi followed by a 12-week online Tai Chi program with easy movements changes blood pressure and cognitive function, focusing on executive function. Then, researchers will test if these changes in heart and brain health are connected, and if they are connected through the changes in brain structure and function. Both the single session and 12-week online Tai Chi program will be practiced by a group of older adults with high blood pressure and normal cognitive function. They will be new to Tai Chi and not exercising regularly.

The hypotheses of the ACTION study are that practicing Tai Chi is good for the heart and brain of older adults with high blood pressure. Specifically, relaxing Tai Chi with gentle movements will reduce blood pressure, and thereby improve cognitive function, particularly executive function.

DETAILED DESCRIPTION:
Hypertension is a major cardiovascular disease risk factor affecting >70% older adults in the United States. It is also a major contributor to cognitive impairment and dementia that affect over 8 million US older adults. Hypertension can cause deteriorations in brain structure and function such as reduced cerebral blood flow, leading to various types of cognitive dysfunction with declines in executive function being the most common. Of note, executive function is a strong predictor of older adults' ability to live independently in the community. Meta-analyses showed that Tai Chi reduces blood pressure (BP) by 12-15 mmHg for systolic BP and 4-6 mmHg for diastolic BP, and improves cognitive function with an effect size of 0.5 for global cognitive function and 0.9 for executive function. Surprisingly, no study has investigated the relationship between the heart and brain health benefits of Tai Chi among older adults with hypertension.

The primary purposes and hypotheses are presented below. Of note, investigators will define the changes of BP, cognitive function focusing on executive function, and brain structure and functions in response to the 12-week online Tai Chi intervention as the chronic change (see primary outcomes 1 to 9).

1. To examine the relationship between the BP and cognitive function, focusing on executive function, response to a 12-wk online Tai Chi intervention. Investigators hypothesize that the BP and cognitive function, focusing on executive function, response to a 12-wk online Tai Chi intervention will be positively correlated.
2. To examine changes in measures of brain structure and functions in response to a 12-wk online Tai Chi intervention, and explore their associations with the BP and cognitive function, focusing on executive function, responses to Tai Chi. Investigators hypothesize that the relationship between the BP and cognitive function, focusing on executive function, responses to the 12-wk online Tai Chi intervention is mediated by the changes in brain structure and function.

The secondary purposes are to examine the relationship between the BP and cognitive function, focusing on executive function, response to a single session of Tai Chi exercise. Investigators hypothesize that the BP and cognitive function, focusing on executive function, response to a single session of Tai Chi exercise will be positively correlated. Of note, investigators will define the changes of BP, cognitive function focusing on executive function in response to a single session of Tai Chi exercise as the acute change (see secondary outcomes 1 to 5).

The participants will be randomized to either a Tai Chi (n=10) or control group (n=10). Participants will receive informed consent material and attend live online Q&A sessions. Participants who signed the informed consent form will attend online visits 1 and 2, and in-person visit 3 to complete eligibility screening. For pre-intervention measures, participants will attend online visit 3 and in-person visits 4 and 5. In-person visits 4 and 5 will be in randomized order and include: 1) the Acute Exercise Visit A during which participants will attend a 45-minute Tai Chi exercise session at the local senior center; and 2) the Control and Magnetic Resonance Imaging [MRI] Visit A at the Brain Imaging Research Center [BIRC] at UConn Storrs during which participants will attend a 45-minute sham control session (i.e., watching Tai Chi themed video). A trained, blinded research assistant will: 1) measure resting BP and cognitive function before and after the 45-minute Tai Chi session in the Acute Exercise Visit A and the 45-minute sham control session in the Control and MRI Visit A; and 2) attach participants to a 24-hour ambulatory BP (ABP) monitor at the end of both the Acute Exercise Visit A and the Control and MRI Visit A that will be worn to the next morning. In addition, participants will participate in an 60-minute MRI scanning session at BIRC in the Control and MRI Visit A. The 12-week online Tai Chi intervention will start after in-person visit 5, participants assigned to the Tai Chi group will attend live online Tai Chi sessions led by a certified Tai Chi instructor for 3 sessions/week, 45 minutes/session for 12 weeks. The participants will also practice Tai Chi at home between sessions using instructional video that will be shared with them at the end of each live online Tai Chi session. Meanwhile, participants in the control group will perform only their regular habitual daily activities throughout the 12-week study. After the 12-week intervention period, participants will attend in-person visit 6 (Control and MRI Visit B) at the BIRC with procedures identical to those conducted in in-person visit 4 or 5 (Control and MRI Visit A). Participants will attend in-person visit 7 (Acute Exercise Visit B) at the local senior center with procedures identical to those conducted in in-person visit 4 or 5 (Acute Exercise Visit A).

ELIGIBILITY:
Inclusion criteria:

* All participants will have established hypertension evidenced by awake ambulatory systolic blood pressure (ASBP)≥130 mmHg or awake ambulatory diastolic blood pressure (ADBP)≥80 or taking antihypertensive medication regardless of the awake ASBP and awake ADBP values. In addition, participants will have blood pressure (BP) within the safe range to exercise evidenced by awake ASBP<145 mmHg and awake ADBP<90 regardless of the use of BP medications.
* For women only, participants need to be postmenopausal evidenced by having experienced >6 consecutive months without menstruation. This is because menstruation could potentially influence BP.
* Participants will be free of Tai Chi practice in the past 12 months
* Participants will, at least, have graduated from high school or have obtained GED.
* Participants will have intact cognitive function evidenced by scoring 25 or higher on the Mini Mental State Examination.
* Participants will be physically inactive as did not exercise for 30 min or more per day at moderate intensity on 3 or more days per week in the past 12 weeks. Subjects will not have physically demanding occupations.
* Participants will consume <2 alcoholic drinks daily because the effects of alcohol may obscure the BP response to exercise.
* Participants will be non-smokers for at least 6 months prior to entry because the effects of tobacco may obscure the BP response to exercise.
* Participants need to have sufficient access to internet and electronic equipment (e.g., laptop, desktop, tablet) to participate in virtual research visits and live online Tai Chi sessions, and email study personnel.

Exclusion criteria:

* Participants will have no contradictions to fully participate in ACTION. They will be excluded if they have: 1) signs or symptoms suggestive of cardiovascular, renal, and metabolic disease; 2) psychiatric and neurological disorders such as general anxiety and depression; 3) body mass index <18.5 kg.m^-2 or >35 Kg·m^-2) orthopedic problems likely to restrict Tai Chi exercise in standing position; 5) contradictions to MRI scans to the brain.
* If the participants has been diagnosed with chronic diseases that require medical clearance to exercise that include cardiovascular, renal, and metabolic disease, the PI and the study medical director will review the participants's medical history and determine if it is safe for him or her to participate in ACTION. If determined unsafe to exercise, the participant will be excluded.
* For participants who have been diagnosed with cancer, only those who have had cancer under remission for 6 months or longer will be considered for inclusion. Otherwise, the participant will be excluded.
* Cancer survivors will be excluded if they: 1) had lung, abdominal surgery, or ostomy within the past 6 months; 2) are currently experiencing ataxia, extreme fatigue, severe nutritional deficiencies, worsening/changing physical condition (i.e., lymphedema exacerbation), bone metastases. For other cancer survivors, the PI and the study medical director will review the participant's medical history and determine if it is safe for him or her to participate in ACTION. If determined unsafe to exercise, the participant will be excluded.
* Participants who have extensive experience with Tai Chi, defined as have practiced Tai Chi for ≥2 sessions/week for ≥3 months continuously, will be excluded.
* Participants who have physically demanding occupations will be excluded.
* Participants acknowledging illicit drug use within the past 5 years will not be recruited.
* Participants taking any medications, except for corticosteroids and hypnotics, should: 1) have been taking the medications for ≥3 months prior to entry; and 2) maintain their routine of taking the medications throughout the study when possible. Otherwise, the participant will be excluded.
* Participants who take corticosteroids and hypnotics as needed will not be recruited because these medications could potentially influence BP and brain blood flow and function.
* Participants taking any nutritional supplements other than a 1-a-day vitamin, cold medications, and herbal supplements would be asked to discontinue these medications before entering the study or be excluded.
* Changes in diet and weight have the potential to obscure and/or augment the influence of our Tai Chi intervention on BP. Participants will be excluded if they are seeking to gain or lose weight or had a weight change of >5 lb in the past 3 months. Investigators will also not recruit subjects unwilling to maintain their habitual diet throughout study participation.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic Change in Resting Systolic and Diastolic Blood Pressure (BP) | Chronic changes in RSBP and RDBP will be calculated as the resting BP at Visit 6 in week 15 (pre-sham control session in Control and MRI Visit B) minus resting BP measured at Visit 4 or 5 in week 2 (pre-sham control session in Control and MRI Visit A).
  Investigators will measure resting systolic BP (RSBP) and resting diastolic BP (RDBP) according to standards set by the American Heart Association using the OMRON automated BP monitors model HEM-705CPN in mmHg.
Chronic Change in Ambulatory Blood Pressure (BP) | Chronic changes in ASBP and ADBP will be calculated as ambulatory BP measured at Visit 6 in week 15 (Control and MRI Visit B) minus the ambulatory BP measured at Visit 4 or 5 in week 2 (Control and MRI Visit A).
  Investigators will measure ambulatory systolic BP (ASBP) and ambulatory diastolic BP (ADBP) with Oscar2 automatic noninvasive ambulatory BP monitor (Suntech Medical Instruments Inc., Raleigh, NC). Ambulatory BP readings will be averaged over hourly intervals for the 'awake', 'sleep', and '24-hour' ambulatory BP in mmHg.
Chronic Change in the Stroop Color and Word Test (SCWT) | Chronic Change in the SCWT will be calculated as SCWT measured at Visit 7 in week 15 (pre-Tai Chi session in the Acute Exercise Visit B) minus the SCWT measured at Visit 4 or 5 in week 2 (pre-Tai Chi session in the Acute Exercise Visit A).
  The SCWT is a validated measurement of executive functions and response inhibition. Participants will be given 45 seconds for each of the three tasks. The trained investigator will count the number of uncorrected errors (i.e., errors without spontaneous corrections from the subject) in each task.response inhibition. Participants will be given 45 seconds for each of the three tasks. The trained investigator will count the number of uncorrected errors (i.e., errors without spontaneous corrections from the subject) in each task.
Chronic Change in the Letter and Category Fluency Test (LCFT) | Chronic Change in the LCFT will be calculated as the LCFT measured at Visit 7 in week 15 (pre-Tai Chi session in the Acute Exercise Visit B) minus the LCFT measured at Visit 4 or 5 in week 2 (pre-Tai Chi session in the Acute Exercise Visit A).
  The LCFT is a validated measurement to assess phonemic and semantic verbal fluency. The number of words in each of the two tasks will be counted by the trained investigator.
Chronic Change in the Hopkins Verbal Learning Test (HVLT) | Chronic change in the HVLT will be calculated as the HVLT measured at Visit 6 in week 15 (pre-sham control session in Control and MRI Visit B) minus the HVLT measured at Visit 4 or 5 in week 2 (pre-sham control session in Control and MRI Visit A).
  The HVLT is a validated measurement to assess verbal learning and memory. All responses (recalled words and yes/no answers) will be recorded by the trained investigator for each of the four tasks. Trained investigators will calculate the raw scores based on total recall, delayed recall, retention (% retained), and a recognition discrimination index.
Chronic Change in the Trial Making Test A and B (TMT) | Chronic change in the TMT will be calculated as the TMT measured at Visit 6 in week 15 (pre-sham control session in Control and MRI Visit B) minus the TMT measured at Visit 4 or 5 in week 2 (pre-sham control session in Control and MRI Visit A).
  The TMT is a two-part validated measurement of executive function and cognitive flexibility. Participants will be allowed up to 180 seconds to complete the TMT A and up to 300 seconds to complete the TMT B. The time to complete each task will yield a raw score in seconds.
Chronic Change in the Computerized California Assessment Package-Abbreviated Version (CalCAP) | Chronic change in the CalCAP will be calculated as the CalCAP measured at Visit 6 in week 15 (pre-sham control session in Control and MRI Visit B) minus the CalCAP measured at Visit 4 or 5 in week 2 (pre-sham control session in Control and MRI Visit A).
  The CalCAP presents a series of brief reaction time tasks designed to assess speeded information processing and psychomotor functioning. Frequency of correct responses to target stimuli will be recorded as true positive responses, and participants' responses to nontarget stimuli will be classified as false positives. The responses will be recorded in milliseconds from the stimulus onset to the manual reaction by the participants.
Chronic Change in the NIH Toolbox Flanker Inhibitory Control and Attention Test (FLANKER) | Chronic change in the FLANKER will be calculated as FLANKER measured at Visit 6 in week 15 (pre-sham control session in Control and MRI Visit B) minus the FLANKER measured at Visit 4 or 5 in week 2 (pre-sham control session in Control and MRI Visit A).
  The FLANKER is a validated measurement of attention and inhibitory control. The adjusted and unadjusted score based on number of correct answers and reaction time will be calculated by the NIH Toolbox automatically.
Chronic Change in Brain Structure and Function measured by Magnetic Resonance Imaging Scans (MRI) | Chronic Change in MRI will be calculated as MRI obtained at Visit 6 in week 15 (Control and MRI Visit B) minus MRI obtained at Visit 4 or 5 in week 1 (Control and MRI Visit A).
  The two MRI scan sessions will be identical and will each take about 60 minutes. Data will be collected on a 3.0 Tesla Siemens Prisma MRI Scanner (Siemens Medical Solutions, Erlangen, Germany) using the body coil for transmission, and a 64-channel phased-array head/neck coil for reception and multi-shell imaging for functional MRI. Specific scans include: 1) T1-weighted 3D magnetization prepared rapid gradient echo (MPRAGE) imaging scan; 2) T2-weighted 3D-Fast Spin Echo, fluid attenuated inversion recovery (FLAIR) imaging scan; 3) task related functional MRI gradient echo-planar imaging (EPI) scan with a block-event mixed design task which includes memory encoding, memory retrieval, and go/no-go distraction blocks; and 4) diffusion tensor imaging (DTI) scan.

SECONDARY OUTCOMES:
Acute Change in Resting Blood Pressure (BP) | Acute changes in RSBP and RDBP will be calculated as (post - pre-Tai Chi session resting BP in the Acute Tai Chi Visit A or B) minus (post - pre-sham control resting BP in the Control and MRI Visit A or B).
  Investigators will measure resting systolic BP (RSBP) and resting diastolic BP (RDBP) according to standards set by the American Heart Association using the OMRON automated BP monitors model HEM-705CPN in mmHg.
Acute Change in Ambulatory Blood Pressure (BP) | Acute changes in ASBP and ADBP will be calculated as (ambulatory BP following the Acute Exercise Session A or B - ambulatory BP following the Control and MRI Visit A or B).
  Investigators will measure ambulatory systolic BP (ASBP) and ambulatory diastolic BP (ADBP) with Oscar2 automatic noninvasive ambulatory BP monitor (Suntech Medical Instruments Inc., Raleigh, NC). Ambulatory BP readings will be averaged over hourly intervals for the 'awake', 'sleep', and '24-hour' ambulatory BP in mmHg.
Acute Change in the Trial Making Test A and B (TMT) | Acute change in the TMT will be calculated as (post - pre-Tai Chi session TMT in Acute Exercise Visit A or B) minus (post - pre-sham control session TMT in Control and MRI Visit A or B).
  The TMT is a two-part validated measurement of executive function and cognitive flexibility. Participants will be allowed up to 180 seconds to complete the TMT A and up to 300 seconds to complete the TMT B. The time to complete each task will yield a raw score in seconds.
Acute Change in the Computerized California Assessment Package-Abbreviated Version (CalCAP) | Acute change in the CalCAP will be calculated as (post - pre-Tai Chi session CalCAP in Acute Exercise Visit A or B) minus (post - pre-sham control session CalCAP in Control and MRI Visit A or B).
  The CalCAP presents a series of brief reaction time tasks designed to assess speeded information processing and psychomotor functioning. Frequency of correct responses to target stimuli will be recorded as true positive responses, and participants' responses to nontarget stimuli will be classified as false positives. The responses will be recorded in milliseconds from the stimulus onset to the manual reaction by the participants.
Acute Change in the NIH Toolbox Flanker Inhibitory Control and Attention Test (FLANKER) | Acute change in the FLANKER will be calculated as (post - pre-Tai Chi session FLANKER in Acute Exercise Visit A or B) minus (post - pre-sham control session FLANKER in Control and MRI Visit A or B).
  The FLANKER is a validated measurement of attention and inhibitory control. The adjusted and unadjusted score based on number of correct answers and reaction time will be calculated by the NIH Toolbox automatically.

CONTACTS AND LOCATIONS:
Overall Officials: Linda S Pescatello, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No